CLINICAL TRIAL: NCT01875692
Title: Culture Versus Genomics: Study of Oropharyngeal and Tracheal Flora in Intubated Patients. Can we Better Understand the Development of Ventilator-Acquired Pneumonia (VAP) and Predict Its Causing Pathogen(s)?
Brief Title: Can we Better Understand the Development of VAP and Eventually Predict and Prevent it?
Status: Completed | Type: Observational
Sponsor: University Hospital, Geneva (Other)
Responsible Party: Principal Investigator, Prof. Jacques SCHRENZEL, Professor, University Hospital, Geneva
Other Study IDs: 12-051
Record Dates: First submitted 2013-03-15; First posted 2013-06-12 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Pneumonia, Ventilator-Associated
Keywords: Metagenomic; Ventilator-Associated Pneumonia (VAP)
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Pathogens of ventilator-associated pneumonia (VAP) come from colonizers of the trachea. The hypothesis of the investigators is that during the first days of intubation, independently of the use of antibiotics, there is a change in the oro-pharyngeal flora leading to the selection of one pathogen in the trachea, that will finally be the cause of VAP.

The investigators designed a prospective study including 300 patients intubated for more than 3 days, with daily analysis of oro-pharyngeal juice and tracheal aspirate by culture and metagenomics, in order to determine if this microbiological surveillance permits:

1. To predict a high risk to develop a VAP in the next 48h and even to predict its agent
2. To better understand the development of VAP by studying the evolution of the "respiratory flora" in the context of intubation

DETAILED DESCRIPTION:
BACKGROUND OF THE STUDY:

The ventilator-associated pneumonia (VAP) is responsible for almost half of infections acquired in intensive care, affecting up to 28% of mechanically ventilated patients with a mortality rate ranging from 25 to 50%. The majority of these VAP originate in the sub-glottic juice that accumulates just above the endotracheal tube cuff. Many preventive measures exist and are applied in this institution, including oropharyngeal aspiration every 4 hours and tracheal aspirates every 8 hours. Currently, these aspirates are simply discarded. However, a French study evaluating the colonization and infection of the respiratory tract of patients with acute respiratory distress syndrome (ARDS) has highlighted that the causative agent of VAP is selected in more than 2/3 of the cases in tracheal aspirates several days before the VAP. This suggest that "microbiological surveillance" of daily aspirates may permit the identification of a selected respiratory pathogen later responsible of VAP.

Parallel to this, the rapid development of genomics has highlighted the role of flora (microbiota) and its link with disease (eg, colitis and intestinal microbiota inflammatory). This area is also emerging in the field of respiratory tract infections, for example in patients with chronic obstructive pulmonary disease (COPD) or asthma. There is no description yet of metagenomics changes in respiratory flora of patients intubated with or without VAP, neither evaluation of the benefits of such an approach in relation to classical microbiology. The investigators believe that studying the respiratory flora of ventilated patients could provide clues to better understand the development of VAP.

METHODOLOGY (plan, inclusion and objectives):

Prospective study of 300 intubated patients recruited during a period of 2 years, in whom tracheal aspirates and oropharyngeal juice collected daily will be analyzed by culture and metagenomics, instead of being simply discarded. The results of these analyzes will be used only for research purposes (culture and metagenomics in parallel).

The main objective is to determine whether daily monitoring of oropharyngeal juice and tracheal aspirates by culture identifies the selection of a pathogen among the colonizing flora, which would be predictive of the onset of VAP in 48-72 hours.

The secondary objectives are to obtain new knowledge on the kinetics of colonization and respiratory infections in intubated patients, compare the advantages and disadvantages of a metagenomic approach compared to culture in this context, and study the influence of antibiotherapy in this context.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalised in the adult ICU of HUG (>18 years old)
* Intubated for < 24 hours
* Expected duration of intubation > 4 days (e.g. neurologic disease)

Exclusion Criteria:

* Patients for whom regular tracheal aspirations cannot not be performed (because of unstable intracranial pressure, for example).
* New antibiotic therapy in the week preceding the intubation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU adult patients intubated in the last 24h for a condition that will probably require more than 3 days of mechanical ventilation.
Sampling Method: Non-Probability Sample
Enrollment: 286 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Percentage of cases where tracheal (same for oropharyngeal) aspirate clearly showing a selection of the same pathogen retrieved later in the bronchoalveolar lavage (BAL), when VAP happens. | After 18 months
  This will provide the sensitivity of tracheal culture to identify correctly the agent of VAP before VAP happens.
Percentage of case where the pathogen selected in tracheal (same for oropharyngeal) aspirate do not correspond to the agent of VAP as identified by BAL. | After 18 months
  Helps to determine the "specificity" of tracheal aspirates to predict the agent of VAP.
Percentage of cases where despite the selection of only one pathogen in tracheal aspirate (same for oropharyngeal) aspirate, the patient did never suffer from VAP | After 18 months
  Helps determining the positive and negative predictive values of tracheal aspirates to predict VAP.
Presence of Ventilator-Associated-Pneumonia (VAP) | After 18 month

SECONDARY OUTCOMES:
Percentage of VAP in the study population | After 18 months
Type of bacteria retrieved on intubation day compared to type of bacteria retrieved after 1 week of intubation | After 18 months
  The investigators expect to find normal oropharyngeal flora on intubation day but Gram negative pathogens after one week, despite the absence of antibiotherapy.
  This will be compared with and without antibiotherapy.
Evolution of metagenomics of oropharyngeal - tracheal aspirates in cases (VAP) and control (no VAP) | After 18 months
  For patients suffering from VAP, metagenomics will also be assessed in the BAL. This will give the investigators some clues on the "respiratory flora" equilibrium and its evolution in cases and control

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Schrenzel, Prof., Principal Investigator — University Hospital, Geneva
Locations (1):
- University Hospital, Geneva, Canton of Geneva, Switzerland